CLINICAL TRIAL: NCT07180173
Title: Retrospective Analysis of Upfront Neck Dissection Before Radiotherapy in Stage N3 Nasopharyngeal Carcinoma
Brief Title: Upfront Neck Dissection Before Radiotherapy in Stage N3 Nasopharyngeal Carcinoma: A Retrospective Study
Status: Active, not recruiting | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CE25786B
Record Dates: First submitted 2025-09-11; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Oncology; Radiology
Keywords: Prognosis; Treatment failure; Nasopharyngeal carcinoma; Intensity-modulated radiotherapy
MeSH Terms: conditions — Neoplasms; Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Salvage Neck Treatment — Salvage neck treatment, including neck dissection with or without re-irradiation and/or systemic therapy, administered to patients with stage N3 nasopharyngeal carcinoma after completion of definitive concurrent chemoradiotherapy (CCRT) or induction chemotherapy followed by radiotherapy/CCRT.

SUMMARY:
This retrospective observational study aims to evaluate the association between neck tumor burden and high-risk imaging features with locoregional recurrence and distant metastasis in patients with stage N3 nasopharyngeal carcinoma, and to explore the potential benefits of neck dissection, with or without re-irradiation or systemic therapy, in improving regional control and survival.

The key questions addressed are whether high N burden and high-risk imaging features are significantly correlated with neck recurrence and distant metastasis, and whether salvage neck treatment (such as neck dissection ± re-irradiation/systemic therapy) can improve regional control and survival outcomes in this high-risk population.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma (NPC), due to its anatomical proximity to the skull base and critical cervical structures, is primarily treated with radiotherapy. However, even with current standard treatments, a subset of patients still develop locoregional failure with poor outcomes. Previous data have shown that the 5-year locoregional control rate for stage IV disease is approximately 80.7%, corresponding to a failure rate of about 20%. Among these, patients with T1-4N3 disease have a lower 3-year distant failure-free survival compared with T4N0-2, indicating that high N stage is associated not only with regional recurrence but also with increased risk of distant metastasis. Based on this, we hypothesize that high nodal burden and high-risk imaging features are significantly associated with cervical recurrence and distant metastasis, and that appropriate and timely salvage treatment to the neck (such as neck dissection with or without re-irradiation/systemic therapy) may improve regional control and survival.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Pathologically confirmed diagnosis of nasopharyngeal carcinoma (NPC).
* Stage IV disease (Tany N3) according to the 8th edition of the AJCC staging system.
* Completion of definitive concurrent chemoradiotherapy (CCRT), or induction chemotherapy (IC) followed by radiotherapy/CCRT.
* Availability of complete clinical imaging and medical records before and after treatment for efficacy and prognostic analysis.

Exclusion Criteria:

* Presence of distant metastasis at initial diagnosis.
* Prior history of treatment for other head and neck malignancies, aside from definitive therapy for NPC (to avoid confounding prognosis).
* Incomplete or prematurely discontinued definitive radiotherapy, resulting in failure to complete the planned curative treatment.
* Lack of complete pathology report, clinical imaging, or treatment records, making effective analysis impossible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients aged 18 years or older with pathologically confirmed nasopharyngeal carcinoma (NPC), staged as Stage IV (Tany N3) according to the 8th edition of the AJCC staging system. All participants have completed definitive concurrent chemoradiotherapy (CCRT) or induction chemotherapy (IC) followed by radiotherapy/CCRT, and have complete clinical imaging and medical records before and after treatment for subsequent efficacy and prognostic analysis. This cohort represents high-risk patients with advanced nodal disease, characterized by increased risks of both locoregional recurrence and distant metastasis, making them suitable for evaluating current treatment outcomes and subsequent management strategies.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2026-09-29 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From completion of primary treatment (CCRT or induction chemotherapy plus RT/CCRT) to disease progression, recurrence, or death from any cause, up to 5 years.
  PFS is defined as the time from treatment completion to the first documented disease progression (locoregional recurrence or distant metastasis) or death, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | From treatment completion to death from any cause, up to 5 years.
  OS is defined as the duration from treatment completion until death from any cause.
Locoregional Recurrence-Free Survival (LRRFS) | From treatment completion to the first occurrence of locoregional recurrence, up to 5 years.
  LRRFS is defined as the time from treatment completion to the first documented local or regional recurrence.
Patterns of Failure | From treatment completion to recurrence/metastasis, up to 5 years.
  Documenting the site and timing of failure (local, regional, distant) based on imaging and pathology reports.
Adverse Events of Salvage Treatment | From initiation of salvage therapy to 90 days post-treatment.
  Acute and late adverse events related to salvage neck dissection, re-irradiation, or systemic therapy, graded according to CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

REFERENCES:
- [Background] Chiang CL, Guo Q, Ng WT, Lin S, Ma TSW, Xu Z, Xiao Y, Li J, Lu T, Choi HCW, Chen W, Chau ESC, Luk PHY, Huang SH, O'Sullivan B, Pan J, Lee AWM. Prognostic Factors for Overall Survival in Nasopharyngeal Cancer and Implication for TNM Staging by UICC: A Systematic Review of the Literature. Front Oncol. 2021 Sep 2;11:703995. doi: 10.3389/fonc.2021.703995. eCollection 2021. PMID 34540670
- [Background] Huang CL, Guo R, Li JY, Xu C, Mao YP, Tian L, Lin AH, Sun Y, Ma J, Tang LL. Nasopharyngeal carcinoma treated with intensity-modulated radiotherapy: clinical outcomes and patterns of failure among subsets of 8th AJCC stage IVa. Eur Radiol. 2020 Feb;30(2):816-822. doi: 10.1007/s00330-019-06500-5. Epub 2019 Oct 24. PMID 31650266